CLINICAL TRIAL: NCT05633628
Title: Periodic Continuous Glucose Monitoring to Support a Person-centered Approach During Diabetes Consultations in Patients With Type 2 Diabetes- A Randomised Controlled Study
Brief Title: Periodic Continuous Glucose Monitoring in Patients With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sophiahemmet University (Other)
Collaborators: Swedish Diabetes Foundation (Unknown); OneTwo Analytics AB (Unknown); Sophiahemmet (Unknown)
Responsible Party: Principal Investigator, Unn-Britt Johansson, Principal Investigator, Professor, Sophiahemmet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Periodic Glucose Insights
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: CGM; Personcentered care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodic CGM- Intervention group (Experimental): The participants in the intervention group will be provided with FreeStyle Libre (Abbott Diabetes Care). Participants wear the sensor and check their glucose level for a period of 28 days (14 days X 2) during week 0-4 and week 10-13.Patient's measurement data from the FreeStyle Libre system will be transferred to the OneTwo Analytics (DDA) analysis tool for an automated analysis and this Insight report will be presented to the participants at visit week 4 (digital) and at visit week 16 (clinical). The diabetes nurse and the patient reviews and discuss trends, patterns, and challenges to support the person's self-management care of their type 2 diabetes. This approach is intended to facilitate communication and patient participation and create the conditions for shared informed decisions and health planning.
  Interventions: Behavioral: Periodic CGM group with data analysis report- Intervention group
- Self-monitoring of blood glucose, SMBG and usual care - Control Group (No Intervention): The participants in the control group perform SMBG testing as usual including fasting, pre- or post-prandial measurements. They also receive usual care which comprises consultation with physician diabetes specialist or diabetes nurse depending on individual health care needs.

INTERVENTIONS:
Behavioral: Periodic CGM group with data analysis report- Intervention group — The patients are also instructed to continue to perform SMBG by finger prick if they experience symptoms of hypo- or hyperglycemia. During visit 0 (baseline) the patients is also instructed about how they can log in to the National Diabetes Register (NDR) to access their own NDR's recorded data and use the diabetes questionnaire.
  Arms: Periodic CGM- Intervention group

SUMMARY:
The aim of this randomised controlled trial is to investigate the effectiveness of periodic CGM (continuous glucose monitoring) to support a person-centered approach versus self-monitoring of blood glucose (SMBG) in adults with type 2 diabetes on glucose control and patient reported outcomes.

DETAILED DESCRIPTION:
This is a 16-week prospective, multicenter, randomised, open-labelled, two-armed study in adults with type 2 diabetes conducted at primary care practices in Sweden.

Periodic CGM group- Intervention group:

The participants in the intervention group will be provided with FreeStyle Libre (Abbott Diabetes Care). Participants wear the sensor and check their glucose level for a period of 28 days (14 days X 2) during week 0-4 and week 10-13.Patient's measurement data from the FreeStyle Libre system 2 will be transferred to the OneTwo Analytics (DDA) analysis tool for an automated analysis and this Insight report will be presented to the participants at visit week 4 (digital) and at visit week 16 (clinical). The diabetes nurse and the patient reviews and discuss trends, patterns, and challenges to support the person's self-care management of their type 2 diabetes. This approach is intended to facilitate communication and patient participation and create the conditions for shared informed decisions and health planning.

Self-monitoring of blood glucose, SMBG and usual care - Control Group The participants in the control group perform SMBG testing as usual including fasting, pre- or post-prandial measurements. They also receive usual care which comprises consultation with physician diabetes specialist or diabetes nurse depending on individual health care needs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years
* Type 2 diabetes with a duration of > 6 months
* HbA1c 45-70 mmol/mol
* Have a smartphone
* Experience of self-monitoring of blood glucose prior to the study start

Exclusion Criteria:

* Prandial insulin
* Pregnancy or planning pregnancy during the study
* Breastfeeding
* Renal disease with estimated glomerular filtration rate (eGFR) <45 mL/ min/1.73 m2
* Active malignancy or under investigation for malignancy
* Severe visual impairment
* Severe skin allergy that inhibits the use of a continuous glucose monitoring device
* Glucocorticoids (systemic)
* Planned or currently using weight reduction medications, programs, or surgery
* Cognitively or psychologically unable to participate and read instructions
* Enrolled in other clinical trials
* Eating disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | change at week 16
  mmol/mol

SECONDARY OUTCOMES:
Percentage of time spent in range (Glucose) | change first 28 days in the study compared with the last 28 days
  3.9-10 mmol/l as analyzed by OneTwo Analytics CE marked Decision support Clinic
Percentage time spent in hyperglycaemia | change first 28 days in the study compared with the last 28 days
  > 10 mmol/L as analyzed by OneTwo Analytics CE marked Decision support Clinic
Percentage time spent in hypoglycaemia | change first 28 days in the study compared with the last 28 days
  < 3.9 mmol/L as analyzed by OneTwo Analytics CE marked Decision support Clinic
Average glucose value | change first 28 days in the study compared with the last 28 days
  mmol/L as analyzed by OneTwo Analytics CE marked Decision support Clinic
Standard deviation for glucose value | change first 28 days in the study compared with the last 28 days
  SD as analyzed by OneTwo Analytics CE marked Decision support Clinic
Percentage time in euglycemia, time in target | change first 28 days in the study compared with the last 28 days
  3.9-8.0 mmol/L as analyzed by OneTwo Analytics CE marked Decision support Clinic
Number of hyperglycemic episodes per day | change first 28 days in the study compared with the last 28 days
  Number of hyperglycemic episodes per day as analyzed by OneTwo Analytics CE marked Decision support Clinic
Number of hypoglycemic episodes per day | change first 28 days in the study compared with the last 28 days
  Number of hypoglycemic episodes per day as analyzed by OneTwo Analytics CE marked Decision support Clinic
Data availability in % of all time | change first 28 days in the study compared with the last 28 days
  Data availability in % of all time as analyzed by OneTwo Analytics CE marked Decision support Clinic
Prandial delta within 2 hours, post - pre-prandial values for breakfast, lunch and dinner. | change first 28 days in the study compared with the last 28 days
  Prandial delta within 2 hours, post - pre-prandial values for breakfast, lunch and dinner as analyzed by OneTwo Analytics CE marked Decision support Clinic
Postprandial peak during 2 hours for breakfast, lunch and dinner. | change first 28 days in the study compared with the last 28 days
  Postprandial peak during 2 hours for breakfast, lunch and dinner as analyzed by OneTwo Analytics CE marked Decision support Clinic
Night-time insulin effect | change first 28 days in the study compared with the last 28 days
  Night-time insulin effect as analyzed by OneTwo Analytics CE marked Decision support Clinic
Fasting glucose level | change first 28 days in the study compared with the last 28 days
  Fasting glucose level as analyzed by OneTwo Analytics CE marked Decision support Clinic
The Diabetes Treatment Satisfaction questionnaire | change at week 16
  Includes eight items related to the diabetes treatment over the past weeks.
WHO-5 Well-Being Index | change at week 16
  Brief well-being questionnaire with five items in relation to previous 2 weeks
The Patient Preferences for Patient Participation (4Ps) | change at week 16
  The 4Ps is a questionnaire including 12 items comprising patient´s preferences as well as experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Unn-Britt Johansson, Principal Investigator — Sophiahemmet University
Locations (1):
- Sophiahemmet University, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No